CLINICAL TRIAL: NCT02035202
Title: Real-Time Mobile Cognitive Behavioral Intervention for Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Colin Depp, Associate Professor of Psychiatry, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R01MH100417 (NIH)
Record Dates: First submitted 2013-10-09; First posted 2014-01-14 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2019-08-13 (Actual); Status verified 2019-07

CONDITIONS: Schizophrenia; Bipolar Disorder
MeSH Terms: conditions — Schizophrenia; Bipolar Disorder

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- CBT2go (Experimental): Participants assigned to this condition will attend one session with a therapist to identify cognitive and behavioral strategies around four areas: 1) mood/psychotic symptoms, 2) medication adherence, 3) socialization, and 4) relapse prevention. Subsequently they will answer questions on a mobile device (smartphone) 3 times per day for 12 weeks, and they will receive personalized cognitive and behavioral strategies linked to their momentary responses with bi-monthly telephone support.
  Interventions: Behavioral: CBT2go; Device: Smartphone
- EMA-only (Active Comparator): Participants assigned to this condition will answer questions on a mobile device (smartphone) 3 times per day for 12 weeks but will not receive personalized cognitive and behavioral strategies.
  Interventions: Device: Smartphone
- Standard Care (No Intervention): Participants assigned to this condition will only participate in the assessments.

INTERVENTIONS:
Behavioral: CBT2go — CBT administered using mobile intervention.
  Arms: CBT2go
Device: Smartphone — A smartphone platform will be used to deliver the CBT2go behavioral intervention and the surveys in the EMA-only arm.
  Arms: CBT2go; EMA-only

SUMMARY:
The purpose of this study is to evaluate the effectiveness of a mobile real-time cognitive behavioral intervention for serious mental illness (SMI) and to identify the facilitators, barriers, and costs of implementation. We would like to determine whether the addition of a mobile phone monitoring software program to a brief behavioral intervention for bipolar disorder or schizophrenia improves symptoms arising from the disorders. In this study we will be assessing the feasibility, acceptability and short term effect of the mobile phone enhanced intervention for bipolar disorder and schizophrenia.

DETAILED DESCRIPTION:
Bipolar disorder (BD) and Schizophrenia (SZ) are leading causes of disability and are the costliest disorders to treat among serious mental illnesses. Ample evidence exists that evidence-based psychotherapies such as cognitive behavioral therapy (CBT) produce clinically significant improvements in symptoms of BD and SZ, and yet only 5% of patients in the community can access these treatments. Access to CBT for serious mental illnesses is limited by the restricted pool of trained providers, the resource intensity of these treatments, and cessation of reimbursement for psychological services in many public mental health systems. Our research in BD and SZ over the past five years indicates that mobile phones can provide automated yet personalized cognitive behavioral intervention that is feasible, acceptable, and associated with improvements in symptoms, medication adherence and socialization. Our intervention, called CBT2go, integrates ecological momentary assessment with personalized interventions delivered in the moment that symptoms and related experiences occur. We have developed an innovative platform that functions on various screen types, operating system, or data access technologies, and we have begun to incorporate innovative features into CBT2go, including location-based data and personalized predictive modeling, that can potentially lead to transformative mobile interventions. We propose a research study with the overarching aims of evaluating the effectiveness of CBT2go, gathering necessary data to refine its innovative features, and examining its costs, facilitators, and barriers to implementation in a public mental health system. We propose a randomized controlled trial with three arms: 1) CBT2go, 2) an ecological momentary assessment only condition to control for self-monitoring and device contact, and 3) standard care. A total of 255 participants with either BD or SZ will be recruited from a large public mental health system that has minimal access to CBT. Participants will be assessed at baseline, 6 weeks (mid-treatment), 12 weeks (post-treatment) and 24 weeks (follow-up). The primary outcome of the study will be clinician rated global psychopathology, and secondary outcomes will include medication adherence, social functioning, and mental health service utilization. Recognizing that not all participants will benefit, we propose to examine differential effectiveness in sub-groups. We will also examine mechanisms of change to inform mobile intervention design, focusing on the impact of CBT2go on cognitive insight and dysfunctional attitudes, which are two mediators of change in traditionally delivered CBT. Drawing from experience in implementation research, we will employ a mixed methods approach to assessing the facilitators, barriers, and costs of adoption of CBT2go from perspectives of consumers, technology experts, administrators and front-line clinicians. This study will lay the groundwork for CBT2go to be adapted and implemented with high fidelity in healthcare settings.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female age 18-55
2. MINI Diagnosis of either BD I, SZ, or schizoaffective disorder
3. Currently outpatient, participating in routine psychiatric care and prescribed medications for prior past six months
4. No psychotropic medication changes in the past 3 months
5. Capable of providing signed informed consent

Exclusion Criteria:

1. Diagnosis of dementia, seizure disorder, mental retardation, or past head trauma with loss of consciousness for greater than 20 minutes
2. Cannot complete the assessment battery
3. Visual acuity (Snellen chart), reading ability, and manual dexterity sufficient to navigate a touch screen device
4. Symptoms are in "remission" (i.e, scores on all key BPRS items < 3)
5. Currently participating in any other psychosocial interventions

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 255 (Actual)
Dates: Start 2013-10; Primary Completion 2017-05 (Actual); Study Completion 2017-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Colin Depp, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- UCSD, San Diego, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CBT2go | EMA-only | Standard Care
Started | 85 | 85 | 85
Completed | 77 | 69 | 83
Not Completed | 8 | 16 | 2
Not completed — Lost to Follow-up | 8 | 16 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CBT2go | EMA-only | Standard Care | Total
Number analyzed (Participants) | 77 | 69 | 83 | 229
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 77 | 69 | 83 | 229
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: YEARS] | 51.2 (11.5) | 49.4 (11.1) | 48.1 (11.7) | 49.3 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 28 | 36 | 100
  Male | 41 | 41 | 47 | 129
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 4 | 6 | 5 | 15
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 12 | 17 | 14 | 43
  White | 59 | 45 | 64 | 168
  More than one race | 2 | 0 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 77 | 69 | 83 | 229
Brief Psychiatric Rating Scale TOTAL [Mean (Standard Deviation); unit: units on a scale] — The BPRS-24 includes 24 items that cover depression, anxiety, mania, suicidality, delusions/hallucinations, and unusual behavior. The BPRS is reliable, valid, and sensitive to change in both bipolar disorder and schizophrenia, and therefore enables the examination of diagnosis as a moderator of treatment effect. Twenty four items are rated on a 1-7 scale from present to severe, and the Total Score will be the primary outcome for analyses. It is clinician rated and the minimum score is 24 and the maximum score is 148 and higher scores reflect worse outcome.
  units on a scale | 43.2 (9.7) | 41.6 (11.5) | 42.0 (10.9) | 42.3 (10.7)

OUTCOME MEASURES:

1. Primary Outcome: Score on the Brief Psychiatric Rating Scale (BPRS)
Description: The BPRS-24 includes 24 items that cover depression, anxiety, mania, suicidality, delusions/hallucinations, and unusual behavior. The BPRS is reliable, valid, and sensitive to change in both bipolar disorder and schizophrenia, and therefore enables the examination of diagnosis as a moderator of treatment effect. Twenty four items are rated on a 1-7 scale from present to severe, and the Total Score will be the primary outcome for analyses. It is clinician rated and the minimum score is 24 and the maximum score is 148 and higher scores reflect worse outcome.
Time Frame: Baseline, 6 weeks, 12 weeks, and 24 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT2go | EMA-only | Standard Care
Number analyzed (Participants) | 77 | 69 | 83
units on a scale
  Baseline | 43.2 (9.7) | 41.6 (11.5) | 42.0 (10.9)
  6 weeks | 41.0 (11.1) | 39.6 (7.7) | 41.0 (11.3)
  12 weeks | 39.7 (11.9) | 38.6 (9.1) | 41.0 (11.4)
  24 Weeks | 39.7 (11.9) | 37.6 (10.1) | 41.1 (11.4)

2. Secondary Outcome: SPECIFIC LEVEL OF FUNCTION (SLOF)
Description: The SLOF is an interviewer rated measure that addresses community function in serious mental illness, utilizing a best estimate approach in which data is integrated from interviewer, informant, and participant responses. The score ranges from 30 to 150. Higher scores equal greater function.
Time Frame: Baseline, 12 weeks, 24 weeks
Population: There was missing data due to lack of available informants for the SLOF so that the number analyzed is less than that associated with the other measures
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT2go | EMA-only | Standard Care
Number analyzed (Participants) | 71 | 61 | 73
units on a scale
  Baseline | 126.9 (15.2) | 128.4 (15.51) | 126.9 (16.1)
  12 weeks | 129.1 (15.8) | 127.8 (16.1) | 123.4 (15.8)
  24 Weeks | 130.0 (16.9) | 128.7 (16.3) | 123.3 (18.0)

3. Other Pre Specified Outcome: Dysfunctional Attitudes Scale (DAS)
Description: The DAS is a 40-item self-report subscale indexing maladaptive attitudes, particularly one's ability to perform tasks and one's need for approval from others. The DAS consists of 40 items and each item consists of a statement and each is rated on a 7-point Likert scale (7 = fully agree; 1 = fully disagree). Ten items are reverse coded (items: 2, 6, 12, 17, 24, 29, 30, 35, 37 and 40). The total score is the sum of the 40-items and the range of scores is 40-280, with higher scores indicating more dysfunctional attitudes.
Time Frame: Baseline, mid-point (6 weeks), at post-treatment (12 weeks), 24 week follow up
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT2go | EMA-only | Standard Care
Number analyzed (Participants) | 75 | 62 | 74
units on a scale
  Baseline | 49.9 (18.8) | 49.9 (18.2) | 49.3 (17.8)
  6 weels | 47.8 (19.0) | 49.9 (18.0) | 49.6 (15.4)
  12 weeks | 47.0 (18.3) | 46.0 (17.4) | 51.3 (18.9)
  24 weeks | 45.2 (19.0) | 48.0 (19) | 48.6 (16.4)

ADVERSE EVENTS:
Time Frame: 6 months
Description: Adverse event: Any unfavorable and unintended sign, symptom or disease temporally associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure.
  Serious Adverse Event: Any AE that results in any of the following outcomes:
  * Death
  * Life-threatening event requiring inpatient hospitalization or prolongation of existing hospitalization
  * Persistent or significant disability/incapacity
Arm/Group | CBT2go | EMA-only | Standard Care
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/85 | 0/85
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/85 | 0/85
Other Adverse Events (participants affected / at risk) | 10/85 | 12/85 | 9/85
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CBT2go (N=85) | EMA-only (N=85) | Standard Care (N=85)
Hospitalization (Psychiatric disorders) | 10 (10) | 12 (12) | 9 (9)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-05-17): https://cdn.clinicaltrials.gov/large-docs/02/NCT02035202/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-01): https://cdn.clinicaltrials.gov/large-docs/02/NCT02035202/SAP_001.pdf